CLINICAL TRIAL: NCT03803969
Title: ConfirmRxTM: Effects of Patient Posture and Physical Activity
Brief Title: ConfirmRxTM: Posture and Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ABT-CIP-10250 Ver. A.1
Record Dates: First submitted 2019-01-10; First posted 2019-01-15 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Syncope; Cryptogenic Stroke
Keywords: Syncope; Cryptogenic Stroke; Physical activity; Posture
MeSH Terms: conditions — Syncope; Ischemic Stroke; Motor Activity

STUDY DESIGN:
Intervention Model Description: This is a prospective, single arm, unblinded, non-randomized, open-label, multi-center, post-market clinical investigation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ConfirmRx (Insertable Cardiac Monitor) (Other): This is a single arm study where in patients with an approved indication for a cardiac monitor will receive a ConfirmRx Device.
  Interventions: Device: ConfirmRx (Insertable Cardiac Monitor)

INTERVENTIONS:
Device: ConfirmRx (Insertable Cardiac Monitor) — This study is designed to characterise the safety and performance of the ConfirmRx device by assessing quality of signal attained from the device with changes in posture and physical activity at implant and 30days post procedure. The study is also intended to assess gross migrations of the device at 30days post implant.

SUMMARY:
Insertable Cardiac Monitor's (ICM's) such as Confirm Rx™ are leadless devices implanted for long-term heart rhythm monitoring in the diagnosis and management of clinical conditions such as recurrent unexplained syncope, cryptogenic stroke, ventricular arrhythmias and monitoring atrial fibrillations (AF) post ablation. There is limited data on variations seen in signal sensing with changes in physical activity and posture. This single arm, non-randomized, open-label, multi-center, clinical investigation of 100 subjects is designed to characterise the safety and performance of Confirm RxTM by assessing quality of signal attained from the device with changes in posture and physical activity at implant and 30days post procedure. The study is also intended to assess gross migrations of the device at 30days post implant.

DETAILED DESCRIPTION:
Syncope is a condition that has vexed cardiologists worldwide due to its elusive nature. Often a third of patients with syncope remain undiagnosed despite assessments by multidisciplinary teams and the availability of various screening techniques such as electrocardiography, 24-h Holter monitoring, carotid sinus massage, echocardiography, exercise testing, head-up tilt test, and electrophysiological studies. Recently, ICM's have been developed to continuously monitor heart rhythm and thus aid in the diagnoses and management of clinical conditions such as ventricular arrhythmias, cryptogenic stroke, recurrent unexplained syncope and for monitoring atrial fibrillations (AF) post ablation. ICM's such as Confirm Rx from Abbott are leadless devices that detect arrhythmias largely depending on sensing of changes in R-R interval and R wave amplitude in the ECG signal. Whilst ICM's have been helpful in detecting arrhythmias in up to 40% of these patients with unexplained syncope, there is paucity of data regarding changes in signal quality with variations in body posture, physical activity and device movements that could potentially have effects on ECG signal and thus event detection. To this extent, this is an Abbott sponsored prospective, single arm, non-randomized, open-label, multi-center, clinical trial of 100 subjects designed to characterize the safety and performance of Confirm Rx™ in relation to physical activity and posture in these subjects with unexplained syncope.

ConfirmRx™ has come a long way since its inception with a significant reduction in size (78% reduction by volume) that has led to relatively simple insertion procedures through a small skin incision. The less complicated insertion process permits the insertion procedure to take place in settings besides operating rooms and furthermore, smaller devices are associated with significantly lower incidence of infections. We believe that this study will add to growing body of evidence of the efficacy of ConfirmRx.

The primary objective of this clinical investigation is to characterise the safety and performance of the Confirm Rx™ Insertable Cardiac Monitor (ICM) by assessing quality of signal attained from device post implant with changes in posture and physical activity at implant and 30days post procedure.

Primary Endpoints

* Changes in R-wave amplitudes at time of insertion and 30 days post-insertion.
* Changes in R-wave amplitude with below defined movements at time of insertion, and 30days post-insertion.

To identify any gross migration of Confirm Rx device 30 days following implant. Secondary Endpoints

* Change in measured distance/position of scar relative to distance from left lateral sternal border at baseline and 30 days
* Measurement of tip of device from left lateral sternal border
* Deviation of proximal tip of device from scar compared to baseline

ELIGIBILITY:
Inclusion Criteria:

Eligible patients will meet all the following:

1. Subjects are 18 years of age or older, or of legal age to give informed consent specific to state and national law.
2. Subject must provide written informed consent prior to any clinical investigation related procedure.
3. Have an approved indication for continuous arrhythmia monitoring with an Insertable Cardiac Monitor.
4. Should be willing and able to comply with the prescribed follow-up tests and schedule of evaluations.
5. Female subjects of child-bearing potential should have a negative pregnancy test done within 7 days prior to the index procedure per site standard test.

Exclusion Criteria:

Patients will be excluded if they meet any of the following:

1. Subject has previously received an Insertable Cardiac Monitor.
2. Subject is currently enrolled or intend to participate in another clinical investigation, which could confound the results of this trial during this clinical study as determined by the sponsor.
3. Pregnant or nursing subjects and those who plan pregnancy during the clinical investigation follow-up period.
4. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Characterisation of the safety and performance of Confirm Rx™ with changes in posture and physical activity at implant and 30days post procedure | 30+15 days post procedure
  Patient performs defined movements post insertion of device and assessments are made on the Merlin Programmer. These are repeated 30+15 days post procedure

SECONDARY OUTCOMES:
Identification of any gross migration of Confirm Rx device 30 days following implant | 30+15 days post procedure
  Measurements of location of the device is recorded post procedure and then measured again 30+15 days post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Pavia, MBBS, FRACP, Principal Investigator — Fundacion GenesisCare
Locations (8):
- Australia (8):
  - The Wesley Hospital, Auchenflower, Queensland
  - Friendly Society Private Hospital, Bundaberg, Queensland
  - Greenslopes Private Hospital, Greenslopes, Queensland
  - St Andrews Hospital, Adelaide, South Australia
  - Warringal Private Hospital, Heidelberg, Victoria
  - The Valley Private Hospital, Mulgrave, Victoria
  - St John of God Murdoch Hospital, Murdoch, Western Australia
  - Mount Hospital, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Swale M, Paul V, Delacroix S, Young G, McSpadden L, Ryu K, Di Fiore D, Santos M, Tan I, Conradie A, Duong M, Schwarz N, Worthley S, Pavia S. Changes in R-wave amplitude at implantation are associated with gender and orientation of insertable cardiac monitor: observations from the confirm Rx body posture and physical activity study. BMC Cardiovasc Disord. 2022 Oct 8;22(1):439. doi: 10.1186/s12872-022-02752-0. PMID 36209063